CLINICAL TRIAL: NCT05345548
Title: Sensitivity, Threshold, Tolerance and Pain Recognition in Schizophrenia Patients and Their Relatives
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Einat Mader, Principal Investigator, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0041-19-EMC
Record Dates: First submitted 2022-03-14; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Pain Recognition; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cold Pressor test (Experimental)
  Interventions: Diagnostic Test: Cold Pressor test

INTERVENTIONS:
Diagnostic Test: Cold Pressor test — Cold Pressor test will be done for 3 minute duration maximum

SUMMARY:
It has been known that schizophrenia patients have a reduced ability to recognize both their own pain and the pain of others. The patients' pain judgement is not correlated with their affective or cognitive empathic capacities. These results suggest that changes in pain recognition in schizophrenia patients reflect specific dysfunctions in pain processing .

Schizophrenia patients have a reduced ability to recognize both their own pain. This deficit is not related to their empathic capacities . The correlation between pain perception in schizophrenia patients and their ability to evaluate their own pain is still unknown.

Pain insensitivity to pressure has been described in the context of schizophrenic illness was also evident in the biological relatives of those with the disorder. It is still unclear whether relatives of schizophrenia patients have aberrations in assessing their own pain in different imaginary situations.

Animal models are important tools in the study of psychiatric disorders and the mechanism of action of antipsychotic and other psychiatric drugs. Positive symptoms of schizophrenia are difficult to model in rodents, but locomotor hyperactivity in response to a novel environment were reported as correlated with positive symptoms . On the other hand, negative symptoms such as social interaction and anhedonia and cognitive processing (e.g. emotional memory, sensorimotor gating, and associative learning) can be investigated in animal models with a high degree of validity . Furthermore, in most schizophrenia-like animal models, both first and second-generation antipsychotic drugs are reported to be effective in ameliorating behavioral abnormalities.

It is well establish that patients with schizophrenia have been shown to display decreased sensitivity to pain, and antipsychotics are used to treat chronic pain. For example, chronic administration of phencyclidine or ketamine, psychomimetic drugs, produces decreased sensitivity to mechanical stimulation, and increased pain tolerance. The classic antipsychotic drug fluphenazine has anti-allodynic properties in multiple rodent models of nerve injury-induced neuropathic pain. An analgesic effect of quetiapine in the Cancer-induced bone pain animal model have been demonstrated. However, the mechanism of action to relive pain is still under debate and may differ between different agents. Animal models of acute and chronic pain allow evaluating the effects of analgesics drugs and other components on pain sensation and transmission, and underlining their molecular mechanism. Usually, these tests rely on an escape behavior or a withdrawal reflex as an index of pain. One known method of measuring responses to thermal stimuli involves application of a noxious thermal stimulus (hot or cold). This method has been used in order to investigate new analgesic components.

Study hypothesis Schizophrenia patients and their biological relatives who have an aberrant sensation of pain also have a reduced capability to evaluate their own pain.

Primary objectives

1. Demonstrate that schizophrenia patients who suffer from pain insensitivity also have a reduced capability to evaluate their own pain, compared to population without a mental illness.
2. Prove that the severity of pain insensitivity in schizophrenia patients is correlated to the degree of their ability to assess their own pain in different imaginary situations.

Secondary objective

1. Demonstrate that healthy biological relatives of schizophrenia patients have aberrations in assessing their own pain.
2. Find the correlation between pain insensitivity in schizophrenia patients to pain insensitivity in their relatives.
3. Find the correlation between the degrees in pain recognition in schizophrenia patients to pain recognition in their biological relatives.
4. Investigate the impact of anti-psychotic drugs on pain threshold of schizophrenia patients.

Study design This study is a prospective cross-sectional trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must meet DSM-5 criteria for a diagnosis of schizophrenia.
2. Patients above 18 years of age.
3. Sufficient knowledge of the Hebrew language
4. A stabled mental state. If hospitalized, patients are scheduled for discharge on the basis of clinical assessment of psychiatric symptoms.

Exclusion Criteria:

1. Mental co-morbidity.
2. Peripheral neuropathies, upper limb trauma, chronic pain conditions.
3. Alcohol or drug use.
4. Usage of any pain reliever medications during the week before recruitment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-29 (Actual); Primary Completion 2023-12-29 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Schizophrenia patients and their biological relatives who have an aberrant sensation of pain also have a reduced capability to evaluate their own pain. | 20 minutes
  severity of pain insensitivity in schizophrenia patients is correlated to the degree of their ability to assess their own pain in different imaginary situations.using pain sensitivity questionnaire & cold pressor test

CONTACTS AND LOCATIONS:
Overall Officials: Einat Mader, MD, Principal Investigator — haemek medical center
Locations (1):
- Haemek medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No